CLINICAL TRIAL: NCT07028658
Title: Efficacité de la rééducation Orthophonique de la Lecture Labiale Des Patients appareillés Auditifs : étude SCED
Brief Title: Effectiveness of Speech Therapy for Lip-reading in Patients With Hearing Aids: SCED Study
Acronym: SCEDuLL
Status: Not yet recruiting | Type: Observational
Sponsor: Institut Pasteur (Industry)
Collaborators: IHU reConnect (Unknown)
Responsible Party: Sponsor
Other Study IDs: 2024-135_SCEDuLL; 2025-A00506-23 (Other: ID-RCB)
Record Dates: First submitted 2025-06-11; First posted 2025-06-19 (Actual); Last update posted 2025-06-19 (Actual); Status verified 2025-06

CONDITIONS: Hearing Loss, Bilateral or Unilateral
MeSH Terms: conditions — Hearing Loss

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Speechreading training — The patient will undergo 16 lip reading training sessions. By developing functional lip reading skills, they will be able to fill in the gaps in auditory information they miss, especially in loud or noisy settings

SUMMARY:
This study aims to investigate whether lip reading rehabilitation improves viseme recognition in individuals with hearing impairments who use hearing aids.

ELIGIBILITY:
Inclusion Criteria:

* Patient aged 18 or older
* Affiliated with a social security system
* Moderate to severe bilateral post-lingual hearing loss, fitted with hearing aids for more than 6 months
* Wearing hearing aids for a minimum of 8 hours/day on average over the past month
* Intelligibility in quiet > 80% correct responses at 60 dB (Lafon cochlear list)
* Difficulty in noisy environments rated > 6 on a 0-10 EVA scale
* French language comprehension level of at least B1 CEFR (Common European Framework of Reference for Languages)
* Willing to participate in speech therapy rehabilitation at a rate of 2 sessions per week

Exclusion Criteria:

* Patient who has already undergone speech therapy rehabilitation as part of their hearing loss treatment
* Diagnosis of neurodegenerative disease or history of brain injury (traumatic brain injury, stroke, tumor, meningitis, etc.)
* Uncorrected vision or visual impairment affecting lip reading (e.g. AMD, glaucoma, unoperated cataract, etc.)
* Presence of severe tinnitus (score > 56) on the Tinnitus Handicap Inventory (THI) questionnaire
* Significant cognitive impairment (CODEX C or D) or Montreal Cognitive Assessment (MOCA) score < 23

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population consists of hearing-impaired individuals with hearing aids
Sampling Method: Non-Probability Sample
Enrollment: 8 (Estimated)
Dates: Start 2025-09 (Estimated); Primary Completion 2026-09 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Repetition score, in words (with and without labial doppelganger) of Lafon's cochlear lists presented on video support in visual-only modality | 26 sessions (4,5 months)
Repetition score, in visemes (with and without labial doppelganger) of Lafon's cochlear lists presented on video support in visual-only modality | 26 sessions (4,5 months)

SECONDARY OUTCOMES:
Repetition score of 10 non-words on recorded support with a Signal-to-Noise Ratio of 10 | 26 sessions (4,5 months)
Repetition score of sentences on video support in audiovisual modality | 26 sessions (4,5 months)
Identification score of two sequences of musical notes | 26 sessions (4,5 months)
Impact of speech therapy rehabilitation on quality of life | 26 sessions (4,5 months)
  AVS from 0 to 10

IPD SHARING:
Plan to Share IPD: Undecided